CLINICAL TRIAL: NCT02869425
Title: A Randomized, Double-Blind, Parallel-Group Study to Assess the Effects of Arbaclofen ER Tablets Compared With Placebo on Sperm Parameters in Male Subjects With Multiple Sclerosis
Brief Title: To Assess Effects of Arbaclofen ER Tablets Compared With Placebo on Sperm Parameters in Male Subjects With MS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: suspended due to inability to enroll subjects
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Collaborators: Osmotica Pharmaceutical US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OS440-PKP06
Record Dates: First submitted 2016-08-03; First posted 2016-08-17 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis; Sperm
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arbaclofen ER Tablets (Experimental): AERT 10 mg twice daily (BID) (20 mg/day) for 7 days, followed by AERT 15 mg BID (30 mg/day) for 7 days
  Interventions: Drug: arbaclofen ER Tablets
- Placebo for Arbaclofen ER Tablets (Placebo Comparator): Matching placebo AERT 10 mg twice daily (BID) (20 mg/day) for 7 days, followed by matching placebo AERT 15 mg BID (30 mg/day) for 7 days
  Interventions: Drug: Placebo for arbaclofen ER tablets

INTERVENTIONS:
Drug: arbaclofen ER Tablets — arbaclofen ER tablets, 10 mg, 15 mg, or 20 mg
  Other Names: AERT
  Arms: Arbaclofen ER Tablets
Drug: Placebo for arbaclofen ER tablets — matching placebo tablets to arbaclofen ER tablets 10 mg, 15 mg or 20 mg
  Other Names: Placebo
  Arms: Placebo for Arbaclofen ER Tablets

SUMMARY:
This study is designed to assess the effects of a therapeutic dose of arbaclofen extended release (ER) tablets compared with placebo on human sperm concentration, motility, and morphology in male subjects with multiple sclerosis (MS).

DETAILED DESCRIPTION:
Primary Objective:

The primary safety objective is to assess the effects of arbaclofen ER tablets (AERT) compared with placebo on sperm concentration from baseline to the end of 90 days of treatment in male subjects with MS.

Secondary Objectives:

The secondary safety objectives are to assess:

* The effects of AERT compared with placebo on the following sperm parameters from baseline to the end of 90 days of treatment in male subjects with MS:

  * Semen volume and total sperm count per ejaculate;
  * Sperm motility;
  * Sperm morphology; and
  * Plasma levels of reproductive hormones: Follicle-stimulating hormone (FSH), luteinizing hormone (LH), and total testosterone;
* The recovery of subjects with 50 % decrease in sperm parameters 90 days after the discontinuation of IP; and
* The safety and tolerability of IP.

ELIGIBILITY:
Inclusion Criteria:

* For a subject to be eligible for participation in this study, all of the following criteria must be met at Screening:

  1. Sign an informed consent form (ICF) indicating willingness and ability to participate in the study;
  2. Be male and between 18 to 55 years old, inclusive, at the time of dosing;
  3. Has an established diagnosis of MS for >6 months; subjects with all types of MS (relapsing remitting, secondary-progressive, primary-progressive, or neuromyelitis optica) can be enrolled in the study if they meet all other eligibility criteria;
  4. Has spasticity in the extremities that requires daily treatment with anti-spasticity drugs in the judgment of the Investigator;
  5. Is able to have an erection and antegrade ejaculation with or without the use of phosphodiesterase 5 inhibitors (sildenafil, tadalfil, etc.);
  6. The average of each semen parameter (except volume) collected at Screening (Visits 1 and 2) will be calculated to determine if the subject meets the following sperm eligibility criteria:

     1. Semen volume > or equal to 1.5 mL,
     2. Total sperm per ejaculation > or equal to 15 million,
     3. Sperm concentration > or equal to 10 million/mL,
     4. Total sperm motility > or equal to 19%, and
     5. White blood cell count <3 million/mL,
  7. Concomitant use of baclofen is permitted during Screening, but subjects must stop baclofen on the day prior to randomization (Visit 3). All other prohibited concomitant medications (Appendix D) must be discontinued prior to randomization (Visit 3);
  8. If receiving disease-modifying medications, these must have been at a stable dose for at least 3 months prior to randomization;
  9. All other medications, including AMPYRA® (e.g., dalfampridine, fampridine, 4 aminopyridine), must have been at a stable dose for at least 3 months prior to randomization;
  10. Absence of infections, peripheral vascular disease, contractures, advanced arthritis, or other conditions that hinder evaluation of joint movement;
  11. Has a creatinine clearance > or equal to 50 mL/min, as calculated by glomerular filtration rate using the Modification of Diet in Renal Disease formula;
  12. Be able to swallow tablets whole;
  13. Be willing to abstain from ejaculation for at least 3 days prior to the collection of each semen sample;
  14. Subject and female partners must agree to use a birth control method while on IP and until 30 days following the last administration of IP; and
  15. If acquisition of a semen sample requires participation of the subject's partner, that partner must sign an informed consent and agree to participate in the study.

Exclusion Criteria:

* Subjects will NOT be eligible for inclusion in the study if any of the following criteria apply:

  1. Had an acute MS exacerbation requiring treatment within 6 weeks of Screening;
  2. Has used intravenous methylprednisolone, or equivalent, within 6 weeks before Visit 1;
  3. Use of concomitant medications that would potentially interfere with the actions of the IP or results of the outcome variables (Appendix D) must be stopped prior to randomization. However, concomitant use of baclofen is permitted during Screening, but subjects must stop baclofen on the day prior to randomization (Visit 3). All other prohibited concomitant medications (Appendix D) must be discontinued prior to randomization (Visit 3);
  4. Has other known reproductive disorders or an identifiable history of infertility:

     1. Vasoligation (surgical ligation of the vas deferens as a means of sterilization);
     2. Azoospermia or severe oligospermia, asthenospermia, teratospermia, leukocytospermia, or any combination of these at baseline; or
     3. Retrograde ejaculation;
  5. Has had a sexually transmitted disease within the last year;
  6. Has severe spasticity that makes the use of placebo medication inappropriate in the judgment of the Investigator;
  7. Has had radiation to the pelvic or groin area;
  8. Has a condition that affects spermatogenesis, such as recent severe genitourinary infections and prostatitis;
  9. Has had previous prostate surgery or vasectomy;
  10. Has been diagnosed by a urologist with any one of the following diseases:

      1. Hydrocele of the tunica vaginalis;
      2. Hematocele;
      3. Torsion of the spermatic cord;
      4. Torsion of the testicular appendage;
      5. Varicocele II or more severe seminal vesiculitis;
      6. Gangrene on the skin of the scrotum;
      7. Cryptorchidism, small testis (12 mL, testicular volumes were determined by use of a Prader orchidometer);
      8. Congenital absence of the vas deferens;
      9. Tuberculosis of the epididymis; or
      10. Chronic prostatitis, defined as > or equal to 3 million/mL white blood cell count in semen samples;
  11. Has a history of unstable psychiatric disease, or current signs and symptoms of significant medical disorders, such as severe, progressive, or uncontrolled pulmonary, cardiac, gastrointestinal, hepatic, renal, genitourinary, hematological, endocrine, immunologic, or neurological disease;
  12. Exhibits suicidality defined as active suicidal plan/intent or active suicidal thoughts in the 6 months before Screening as defined by a suicidal ideation score > or equal to 3 on the C-SSRS, (Appendix B; Has a history of suicide attempts or suicidal ideation within 1 year of Screening as determined by the C-SSRS or medical history or currently is at a serious suicidal risk in the judgment of the Investigator);
  13. Has seizure disorder;
  14. Has significant cognitive deficit, severe or untreated anxiety, or severe or untreated depression, which in the judgment of the Investigator, may interfere with the ability of the subject to participate in the study;
  15. Has a current malignancy or history of malignancy in the last 5 years, except effectively treated basal cell skin carcinoma;
  16. Has advanced or uncontrolled diabetes, human immunodeficiency virus infection, history of hepatitis C or active hepatitis B, or any other significant disease, disorder, or significant laboratory finding which, in the judgment of the Investigator, would put the subject at risk because of participation in the study, influence the result of the study, or affect the subject's ability to participate in the study;
  17. Has planned elective surgery or other procedures requiring general anesthesia during the study;
  18. Current chronic use of long-acting opioids or daily use of short-acting opioids for the treatment of pain;
  19. Has participated in another interventional trial within 30 days of Screening;
  20. Has a positive laboratory test result for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C, or controlled substances; or
  21. Has a history of alcohol dependence, substance abuse, or binge drinking. The subject should avoid heavy drinking during the weeks of sperm sample collection.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-10 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Measure of sperm concentration according to WHO guidelines | 90 days of treatment
  The primary safety objective is to assess the effects of arbaclofen ER tablets (AERT) compared with placebo on sperm concentration from baseline to the end of 90 days of treatment in male subjects with MS. Analyses are performed by World Health Organization (WHO) guidelines (WHO, 2010) to obtain volume (mL), pH, sperm concentration motility, and morphology

SECONDARY OUTCOMES:
Measure of sperm motility according to the WHO guidelines | 90 days of treatment
Measure of Plasma levels of FSH, LH, and total testosterone values and their respective change from baseline values will be summarized by visit | 90 days of treatment
  Plasma levels of FSH, LH, and total testosterone values and their respective change from baseline values will be summarized by visit using an 8-number summary (n, mean, median, SD, 25th percentile, 75th percentile, minimum value, and maximum value).
Measure of Semen volume per ejaculate according to the WHO guidelines | 90 days of treatment
Measure of total sperm count per ejaculate according to the WHO guidelines | 90 days of treatment
Measure of Sperm morphology according to the WHO guidelines | 90 days of treatment
The recovery of subjects with 50% decrease in sperm parameters 90 days after the discontinuation of IP | 90 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kaba, MD, Study Chair — Osmotica Pharmaceutical, VP - Global Clinical Development and Medical Affairs
Locations (2):
- United States (2):
  - Advance Medical Pain Management & Research Clinic, Miami, Florida
  - Meridien Research, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No